CLINICAL TRIAL: NCT00641472
Title: An Evaluation of the Effectiveness of Pulmicort Respules (Budesonide Inhalation Suspension) Versus SINGULAIR (Montelukast Sodium) in Children 2-8 Years Old With Asthma Requiring Controller Therapy.
Brief Title: Pulmicort Respules(Budesonide Inhalation Suspension) vs Singulair, Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Lars-Göran Carlsson
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DX-RES-2103; D5257L00750
Record Dates: First submitted 2008-03-18; First posted 2008-03-24 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: Asthma; Pulmicort; Children; paediatrics; budesonide
MeSH Terms: conditions — Asthma | interventions — Budesonide; montelukast; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Budesonide inhalation suspension
  Interventions: Drug: Budesonide inhalation suspension
- 2 (Active Comparator): Montelukast sodium
  Interventions: Drug: Montelukast Sodium

INTERVENTIONS:
Drug: Budesonide inhalation suspension — 0.5mg
  Other Names: Pulmicort Respules
  Arms: 1
Drug: Montelukast Sodium — 4mg or 5mg
  Other Names: SINGULAR
  Arms: 2

SUMMARY:
A one year study comparing the safety and effectiveness of Pulmicort (0.5mg strength given once a day in the evening) with either 4 or 5mg strength SINGULAR (given once a day in the evening) in children with asthma aged 2 to 8. If allocated to SINGULAR treatment, children aged between 2 and 5 will receive 4mg strength SINGULAR and those aged between 6 and 8 will receive 5mg strength SINGULAR.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 8 at study entry
* At least 3 episodes of wheezing in the previous year that lasted more than 24 hours and affected sleep or symptoms of mild persistent asthma
* use of b-2 agonist treatment on at least 3 of 7 consecutive days or run in

Exclusion Criteria:

* Severe or unstable asthma
* any significant finding at a physical exam
* an exacerbation of asthma in the 30 days before entering the study that might affect study results in judgement of the study doctor

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 380 (Estimated)
Dates: Start 2002-10; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Time to first asthma medication as either step-up PULMICORT RESPULES or oral steroids | Each clinic visit

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events | Each clinic visit
Time to 1st additional asthma medication measured at 12 weeks and 26 weeks | Each clinic visit
Time to 1st acute severe exacerbation (as measured by the need for oral steroids), measured at 12 weeks, 26 weeks, and 52 weeks | Each clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Bertil Andersson, Study Director — AstraZeneca